CLINICAL TRIAL: NCT05552469
Title: A Phase 1b, Open Label, Multi-center, Dose Optimization and Dose Expansion Study to Assess the Safety and Efficacy of DFV890 in Adult Patients With Myeloid Diseases
Brief Title: Dose Optimization and Expansion Study of DFV890 in Adult Patients With Myeloid Diseases
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDFV890G12101; 2022-501406-36-00 (Registry Identifier: EU CTIS)
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Myeloid Diseases
Keywords: MDS; CMML; CCUS; CHRS; NLRP3; Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; inflammasome; CYP2C9
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose escalation: DFV890 low dose (Experimental): DFV890 given as single agent at a low dose
  Interventions: Drug: DFV890
- Dose escalation: DFV890 high dose (Experimental): DFV890 given as single agent at a high dose
  Interventions: Drug: DFV890
- Dose expansion: DFV890 low dose (Experimental): DFV890 given as single agent at a low dose
  Interventions: Drug: DFV890

INTERVENTIONS:
Drug: DFV890 — DFV890 Single Agent

SUMMARY:
Study CDFV890G12101 is an open-label, phase 1b, multicenter study with a randomized two-dose optimization part, and a dose expansion part consisting of three groups evaluating DFV890 in patients with myeloid diseases. The purpose of this study is to assess the safety, tolerability, pharmacokinetics, pharmacodynamics, efficacy and recommended dose for single agent DFV890 in patients with lower risk (LR: very low, low or intermediate risk) myelodysplastic syndromes (LR MDS), lower risk chronic myelomonocytic leukemia (LR CMML) and High-Risk Clonal Cytopenia of Undetermined Significance (HR CCUS).

DETAILED DESCRIPTION:
This research study is to find out if study treatment DFV890 is safe and tolerable, and can help patients who were diagnosed with a myeloid disease such as: very low, low or intermediate risk myelodysplastic syndromes (MDS), very low, low or intermediate risk chronic myelomonocytic leukemia (CMML) and High-Risk Clonal Cytopenia of Undetermined Significance (HR CCUS). The study seeks to determine the optimal dose of DFV890 that is safe and efficacious in patients with myeloid disease. The effectiveness and safety/tolerability of the study treatment is not yet confirmed in this disease setting.

Eligible patients meeting all study entry requirements will be required to provide a sample from their bone marrow at screening and at select study timepoints. All enrolled patients will be dosed for a minimum of twenty-four weeks (6 cycles of treatment) unless they experience side effects related to the study treatment requiring dose interruption/discontinuation, worsening of the disease, and/or if treatment is discontinued at the discretion of the investigator or the patient.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients must be ≥ 18 years of age at the time of signing the informed consent form (ICF) 2. The Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2 3. Patient must be a candidate for serial bone marrow aspirate and/or biopsy according to the institutions guidelines and must be willing to undergo a bone marrow aspirate.

4. Patients must have one of the following for eligibility into the study:

1. In dose optimization: IPSS-R defined very low, low or intermediate risk Myelodysplastic Syndrome (LR MDS) who failed to respond to or did not tolerate ESAs or luspatercept or HMAs and patients with del 5q who failed to respond to or did not tolerate lenalidomide; or
2. In dose optimization and expansion: IPSS-R defined very low, low or intermediate risk Chronic Myelomonocytic Leukemia (LR CMML) who failed to respond to or did not tolerate hydroxyurea or HMAs.
3. changes for dose expansion (applicable as of amendment 3):

   1. LR MDS with ≤ 10% bone marrow blasts, IPSS-R score of ≤ 3.5, transfusion independent (TID) status as per IWG 2006 criteria (requiring <4U pRBC in 8 weeks), clinically meaningful cytopenia(s) and no or limited (<4 months) prior therapy for MDS.
   2. LR CMML patients with symptomatic cytopenias and/or constitutional symptoms refractory, intolerant or unsuitable for standard first-line therapy.
   3. HR-CCUS: Diagnosis of high-risk CCUS by clonal hematopoiesis risk score (CHRS) with clinically meaningful cytopenias and no prior therapy for a myeloid neoplasm.

Key Exclusion Criteria:

1. Systemic antineoplastic therapy (including cytotoxic chemotherapy, alpha-interferon, kinase inhibitors or other targeted small molecules, and toxin-immunoconjugates) or any experimental therapy within 28 days or 5 half-lives, whichever is longer, and recovered from the toxicities before the first dose of study treatment. For patients that received antibodies the washout period is 4 weeks prior to study treatment.

a. For TID LR MDS in Dose Expansion Phase only (applicable as of amendment 03):

1. Prior therapy for MDS administered for >4 months (ESA and luspatercept administered for ≤4 months will be allowed if washout period followed)
2. Concurrent malignancy requiring active systemic therapy
3. Prior or concurrent cytotoxic chemotherapy for MDS at any time

2. History of hypersensitivity to the study treatment or its excipients or to drugs of similar chemical classes.

3. Patients who have previously been treated with agents that have the same mechanism of action as DFV890 as defined in Table 6-7, list of prohibited medications (e.g., drugs targeting the NLRP3 inflammasome pathway and the IL-1 pathway (canakinumab and anakinra)).

4. Use of hematopoietic colony-stimulating growth factors (e.g., G-CSF, GM-CSF, M-CSF), thrombopoietin mimetics or erythroid stimulating agents anytime ≤ 1 week (or 5 half lives, whichever is longer) prior to start of study treatment.

5. Patients receiving:

a. concomitant medications that are known to be modulators of cytochrome P450 enzymes CYP2C9 and/or CYP3A (specifically strong or moderate inducers of CYP2C9, strong inducers of CYP3A enzymes, strong inhibitors of CYP2C9 and/or strong or moderate dual inhibitors of CYP2C9/CYP3A); and b. patients, who are poor CYP2C9 metabolizers receiving concomitant medications known to be strong or moderate inhibitors of CYP3A, whose concomitant medications cannot be discontinued or switched to a different medication within 5 half-lives or 1 week (whichever is longer) prior to start of study treatment and for duration of the study. See Section 6.8 and list of prohibited drugs in Appendix 8 for more details.

6. Dose expansion only: Poor CYP2C9 metabolizers defined as genotype of the CYP2C9 *3/*3 or CYP2C9 *2/*3 allele combinations are excluded.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2027-01-29 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-limiting Toxicities (DLTs) | 28 days
  A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value assessed as clinically relevant, occurring during the DLT monitoring period following the first administration of study treatment.
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 36 months
  Incidence and severity of AEs and SAEs by treatment group, including changes in vital signs, electrocardiograms (ECGs) and laboratory values qualifying and reported as AEs.
Incidence of dose interruptions, discontinuations and reductions | 36 months
  Number of patients with dose adjustments (interruptions, discontinuations and reductions) summarized by treatment group.

SECONDARY OUTCOMES:
Reduction in red blood cell (RBC) / platelet transfusions from baseline for transfusion-dependent (TD) patients | Baseline, 36 months
  The number of red cell or platelet transfusions a patient receives over the course of study treatment will be compared to the patient's baseline transfusion requirements based on the transfusions received during the 16-weeks period prior to the start of study treatment.
Percentage of patients developing transfusion independence (TI) for ≥8 weeks, ≥12 weeks, ≥16 weeks or ≥24 weeks for TD patients | Baseline, 8 weeks, 12 weeks, 16 weeks and 24 weeks
  Percentage of patients who develop red cell or platelet transfusion independence (defined as no red cell or platelet transfusions with a duration lasting for 8, 12, 16, or 24 weeks)
Best overall response (BOR) per 2006 IWG criteria for MDS and CMML | Baseline, 36 months
  BOR is defined as the proportion of patients with best response recorded from the start of the treatment until disease progression/recurrence as per local investigator review and according to 2006 International Working Group (IWG) criteria
Hematological improvement per 2006 IWG criteria for MDS and CMML. | 36 months
  Number of participants with hematologic response will be based on erythroid response (HI-E), platelet response (HI-P), or neutrophil response (HI-N) as per local investigator review and according to 2006 IWG criteria
Rate of hematological improvement per 2006 IWG criteria for CCUS | 36 months
  Rate of hematologic improvement is the proportion of patients with hematologic response based on erythroid response (HI-E), platelet response (HI-P), or neutrophil response (HI-N) as per local investigator review and according to 2006 IWG criteria
Time to onset of transfusion independence | 36 months
  Time to onset of either red cell transfusion independence or platelet transfusion independence
Duration of response (DOR) | 36 months
  DOR is defined as the duration from the first documented onset of any response to the date of progressive disease/relapse or death due to MDS/CMML
Change from baseline in hemoglobin (Hb) | Baseline, 36 months
  Hemoglobin levels over the course of the study will be compared to the patient's baseline to monitor for improvements in anemia
Change from baseline in platelet count | Baseline, 36 months
  Platelet count over the course of the study will be compared to the patient's baseline to monitor for improvements in thrombocytopenia
Change from baseline in Absolute Neutrophil Count/White Blood Cells (ANC/WBC) | Baseline, 36 months
  Ratio ANC/WBC over the course of the study will be compared to the patient's baseline to monitor for improvements in neutropenia
Overall response rate (ORR) for MDS and CMML | 36 months
  ORR is the proportion of patients with a BOR of Complete Remission (CR) or Partial Remission (PR). Response is based on 2006 IWG criteria per local investigator review.
Time to progression to any type of myeloid malignancy (TTPM) for CCUS | 36 months
  TTPM is a time-to-event endpoint that measures the duration from the start of the study to the first documented progression from CCUS to a myeloid neoplasm
Progression free survival (PFS) | 36 months
  PFS is defined as the time from the date of start of treatment to the date of the first documented progression, or death due to any cause. Response is based on 2006 IWG criteria per local investigator review.
Time to progression (TTP) | 36 months
  TTP is defined as the time between date of first documented CR or PR to the date of first documented progression/relapse or death due to any cause, whichever occurs first. Response is based on 2006 IWG criteria per local investigator review.
For CMML: reduction in spleen volume | Baseline, 36 months
  Spleen volume over the course of the study will be compared to the patient's baseline
For CMML: MPN-SAF total symptom score (TSS) | Baseline, 12 months
  The Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) Total Symptom Score (TTS) will be used for the assessment of symptom burden at baseline and monitoring symptom status during the course of treatment. MPN-SAF TSS includes the assessment of 10 symptoms (fatigue, concentration, early satiety, inactivity, night sweats, itching, bone pain, abdominal discomfort, weight loss, and fevers). Severity of each symptom is rated on a 0 (absent/as good as it can be) to 10 (worst-imaginable/as bad as it can be) scale. MPN-SAF TSS has a possible range of scores of 0 to 100 with 100 representing the highest level of symptom severity.
Maximum plasma concentration (Cmax) of DFV890 | 15 days
  Pharmacokinetic parameters will be calculated based on DFV890 plasma concentrations by using non-compartmental method(s). Cmax is defined as the maximum (peak) observed concentration following a dose.
Area under the plasma concentration-time curve from time zero to the last measurable concentration sampling time (AUClast) of DFV890 | 15 days
  Pharmacokinetic parameters will be calculated based on DFV890 plasma concentrations by using non-compartmental method(s). AUClast is defined as the area under the plasma concentration-time curve from time zero to the last measurable concentration sampling time.

CONTACTS AND LOCATIONS:
Locations (28):
- United States (12):
  - Stanford Cancer Center, Stanford, California
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University School of Medicine-Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Sidney Kimmel CCC At JH, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Weill Cornell Medicine NY-Presb, New York, New York
  - Memorial Sloan Kettering Cancer Ctr, New York, New York
  - Vanderbilt University Medical Ctr, Nashville, Tennessee
  - Univ of TX MD Anderson Cancer Cntr, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- France (4):
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
- Germany (4):
  - Novartis Investigative Site, Düsseldorf, North Rhine-Westphalia
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Lübeck
- Novartis Investigative Site, Hong Kong, Hong Kong
- Italy (2):
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Rozzano, MI
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Madrid, Spain
- United Kingdom (3):
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: No